CLINICAL TRIAL: NCT03638388
Title: Rate and Maintenance of Improvement in Myofascial Pain: Dry Needling Alone vs Dry Needling With Intramuscular Electrical Stimulation
Brief Title: Dry Needling vs Dry Needling With ES in Patients With Neck/Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kindyle Brennan (Other)
Responsible Party: Sponsor-Investigator, Kindyle Brennan, Dr. Kindyle L. Brennan, Associate Professor, Doctor of Physical Therapy Program, College of Health Sciences, University of Mary Hardin-Baylor
Organization: University of Mary Hardin-Baylor (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNvDN-ES
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Myofascial Pain; Neck Pain; Shoulder Pain
MeSH Terms: conditions — Neck Pain; Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Experimental There will be two groups in this study, DN alone and DN/IES. Each group will have approximately 22 subjects, resulting in approximately 44 subjects total. Subjects will be randomized into one of the two groups via block randomization method based on order of entry into the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (DN) (Active Comparator): Subjects will receive dry needling treatment, once a week, for 6 weeks.
  Outcomes will be measured at baseline (week 0), 3 weeks after initiation of study (week 3), 6 weeks after initiation of study (week 6), and 6 weeks after last treatment (week 12).
  Interventions: Procedure: Dry needling (DN)
- Dry Needling with Intramuscular electrical stimulation (DNES) (Active Comparator): Subjects will receive dry needling treatment with electrical stimulation, once a week, for 6 weeks.
  Outcomes will be measured at baseline (week 0), 3 weeks after initiation of study (week 3), 6 weeks after initiation of study (week 6), and 6 weeks after last treatment (week 12).
  Interventions: Procedure: Dry needling with intramuscular electrical stimulation (DNES)

INTERVENTIONS:
Procedure: Dry needling (DN) — One to three filament needles (similar to an acupuncture needle) with no medication will be inserted into the tender area of my muscle. The needles will be repositioned a few times to make the muscle twitch. After several twitches occur, the researcher will leave the needles as they are, and the subject will sit in a chair without moving my arms or head, for 10 minutes. After 10 minutes the needles are removed and discarded.
  Arms: Dry Needling (DN)
Procedure: Dry needling with intramuscular electrical stimulation (DNES) — One to three filament needles (similar to an acupuncture needle) with no medication will be inserted into the tender area of the muscle. The needles will be repositioned a few times to make the muscle twitch. After several twitches occur, the researcher will leave the needles as they are, and attach alligator clips to the needles to provide electrical stimulus for 10 minutes while the subject sits in a chair without moving arms or head. After 10 minutes, the electrical stimulus will be turned off and detached, and the needles removed and discarded.
  Arms: Dry Needling with Intramuscular electrical stimulation (DNES)

SUMMARY:
First, we aim to determine if there is a difference in the rate of improvement, as measured by the Neck Disability Index (NDI) and Numerical Pain Rating Scale (NPRS), across a 6 week treatment period between those treated with DN only and those treated with DN and intramuscular electrical stimulation (IES) in subjects with upper trapezius active trigger points (aTrPs). Secondly, we want to determine if improvements in clinical outcomes (NDI and NPRS) of patients with upper trapezius active trigger points (aTrPs) treated with dry needling (DN) alone or dry needling with intramuscular electrical stimulation (DN/IES) are maintained 6 weeks post treatment without further intervention.

Research Questions:

1. Is there a difference in the rate of improvement in NDI and NPRS across a 6 week treatment period in subjects with upper trapezius active trigger points (aTrPs) between those treated with DN only and those treated with DN and intramuscular electrical stimulation (IES)?
2. Are improvements in clinical outcomes (NDI and NPRS) of patients with upper trapezius active trigger points (aTrPs) treated with dry needling (DN) maintained 6 weeks post treatment without further intervention? Tertiary exploration: If improvement is maintained, is there a difference in outcome maintenance between groups? Did improvement increase between 6 and 12 weeks?

ELIGIBILITY:
Inclusion Criteria:

18-59 years old have an active email account have at least one palpable active trigger point (TrP) (located in one or both upper trapezius) English speaking

Exclusion Criteria:

current or previous history of cancer active infection neurologic deficit cognitive deficit pregnancy connective tissue disease and/or autoimmune disorder smoke tobacco received previous DN treatments within 6 weeks of the study, experienced unilateral or bilateral neck/shoulder pain continuously for 3 months or longer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Rate of improvement in numerical pain rating scale between groups | 6 weeks
  Between group difference in within group pain changes
Rate of improvement in Neck Disability Index between groups | 6 weeks
  Between group difference of within group disability changes

SECONDARY OUTCOMES:
Maintenance of pain improvement in both groups | week 6 compared to week 12 data
  Difference between pain scores in both groups between the 6th week of weekly treatment and those 6 weeks after cessation of treatment.
Maintenance of disability improvement in both groups | week 6 compared to week 12 data
  Difference between neck disability scores in both groups between the 6th week of weekly treatment and those 6 weeks after cessation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kindyle L. Brennan, PHD,PT, Principal Investigator — University of Mary Hardin-Baylor
Locations (1):
- University of Mary Hardin-Baylor, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Mayoral-Del Moral O, Sanchez-Sanchez B, Dommerholt J, Gutierrez-Ortega C. Prevalence of Myofascial Pain Syndrome in Chronic Non-Specific Neck Pain: A Population-Based Cross-Sectional Descriptive Study. Pain Med. 2016 Dec;17(12):2369-2377. doi: 10.1093/pm/pnw114. Epub 2016 Jun 20. PMID 28025371
- [Background] Pilgrim J, Engelke Z. Patient Education: Teaching the patient about myofascial pain syndrome. CINAHL Nursing Guide. December 8, 2017;Available from: Nursing Reference Center Plus, Ipswich, MA. Accessed April 13, 2018.
- [Background] Liu L, Huang QM, Liu QG, Ye G, Bo CZ, Chen MJ, Li P. Effectiveness of dry needling for myofascial trigger points associated with neck and shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):944-55. doi: 10.1016/j.apmr.2014.12.015. Epub 2015 Jan 7. PMID 25576642
- [Background] Rock JM, Rainey CE. Treatment of nonspecific thoracic spine pain with trigger point dry needling and intramuscular electrical stimulation: a case series. Int J Sports Phys Ther. 2014 Oct;9(5):699-711. PMID 25328832